CLINICAL TRIAL: NCT02172742
Title: The Effect of BIA 2-093 on the Steady-state Pharmacokinetics of Digoxin in Healthy Volunteers
Brief Title: The Effect of BIA 2-093 on the Steady-state Pharmacokinetics of Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-107
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine acetate; BIA 2-093
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Digoxin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIA 2-093 (Experimental): BIA 2-093 1200 mg (2 tablets 600 mg) ESL, Eslicarbazepine acetate
  Concomitantly with a dose of digoxin (days 1 and 2: loading dose of 0.5 mg/day; days 3 to 8: 0.25 mg/day).
  Interventions: Drug: BIA 2-093; Drug: Digoxin
- Placebo (Placebo Comparator): Placebo (2 tablets matching BIA 2-093 600 mg tablets) PLC, Placebo
  Concomitantly with a dose of digoxin (days 1 and 2: loading dose of 0.5 mg/day; days 3 to 8: 0.25 mg/day).
  Interventions: Drug: Placebo; Drug: Digoxin

INTERVENTIONS:
Drug: BIA 2-093 — BIA 2-093 1200 mg once-daily
  Other Names: ESL, Eslicarbazepine acetate
  Arms: BIA 2-093
Drug: Placebo — matching placebo
  Other Names: PLC, Placebo
  Arms: Placebo
Drug: Digoxin — Digoxin (days 1 and 2: loading dose of 0.5 mg/day; days 3 to 8: 0.25 mg/day).
  Other Names: Lanoxin™

SUMMARY:
The purpose of this study is to investigate the effects of multiple-dose administration of BIA 2-093 on the steady-state pharmacokinetics of digoxin in healthy subjects.

DETAILED DESCRIPTION:
Single centre, multiple-dose, double-blind, randomised, placebo-controlled, two-way crossover study in 12 healthy volunteers. The study consisted of two 8-day treatment periods separated by a washout of 10 or more days. During each of the treatment periods the volunteers received either a daily oral dose of BIA 2-093 1200 mg once-daily (od) or matching placebo, concomitantly with a dose of digoxin (days 1 and 2: loading dose of 0.5 mg/day; days 3 to 8: 0.25 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, neurological examination, and 12-lead ECG.
* Subjects who had clinical laboratory tests clinically acceptable.
* Subjects who were negative for HBs Ag, anti-HCV Ab and anti-HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* In case of female volunteers, subjects who were not of childbearing potential by reason of surgery or, if of childbearing potential, used one of the following methods of contraception: double-barrier or intrauterine device.
* In case of female volunteers, subjects who had a negative pregnancy test at screening.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had any of the following findings on the ECG: QTc interval >440 msec; first-, second- or third-degree atrioventricular block; atrial fibrillation; heart rate below 50 bpm; any other relevant abnormality.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used over the counter medication excluding oral routine vitamins but including mega dose vitamin therapy within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 2 months of their first admission.
* Subjects who had previously received BIA 2-093.
* Subjects who had donated and/or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* In case of female volunteers, subjects who were pregnant or breast-feeding.
* In case of female volunteers, subjects who were of childbearing potential and did not use an authorized effective contraceptive method.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2002-05; Primary Completion 2002-07 (Actual); Study Completion 2002-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz da Silva, MD, PhD, Study Director — Human Pharmacology Unit / BIAL - Portela & Ca, S.A.
Locations (1):
- Human Pharmacology Unit (UFH)Section of Clinical Research (SIC), Department of Research & Development (DID), BIAL - Portela & Cª, SA,, Trofa, Coronado (S.Romão E S. Mamede), Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 2-093 + Placebo: Period 1:
  BIA 2-093 1200 mg with:
  Days 1 and 2: once-daily 0.50 mg digoxin Days 3 to 8: once-daily 0.25 mg odigoxin
  Period 2:
  Placebo with:
  Days 1 and 2: once-daily 0.50 mg digoxin Days 3 to 8: once-daily 0.25 mg odigoxin
- Placebo + BIA 2-093: Period 1:
  Placebo with:
  Days 1 and 2: once-daily 0.50 mg digoxin Days 3 to 8: once-daily 0.25 mg odigoxin
  Period 2:
  BIA 2-093 1200 mg with:
  Days 1 and 2: once-daily 0.50 mg digoxin Days 3 to 8: once-daily 0.25 mg odigoxin
Period: Overall Study
Arm/Group | BIA 2-093 + Placebo | Placebo + BIA 2-093
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 2-093 + Placebo | Placebo + BIA 2-093 | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Steady-state Plasma Concentration
Description: Cmax - Maximum steady-state plasma concentration of BIA 2-005 (BIA 2-093 metabolite) and Digoxin
Time Frame: Day 6 and Day 7: pre-dose; Day 8: pre-dose, ½, 1, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 + Placebo: Both Groups:
  Period 1: BIA 2-093; Period 2: Placebo Period 1: Placebo; Period 2: BIA 2-093
Arm/Group | BIA 2-093 + Placebo
Number analyzed (Participants) | 12
ng/mL
  Cmax (BIA 2-005) | 27571 (8252)
  Cmax (Digoxin) (Digoxin+Placebo) | 2,350 (1,034)
  Cmax (Digoxin) (Digoxin+BIA 2-093) | 1,909 (0,596)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax at Steady-state
Description: Time of Occurrence of Cmax Maximum steady-state plasma concentration of BIA 2-005 (BIA 2-093 metabolite) and Digoxin
Time Frame: Day 6 and Day 7: pre-dose; Day 8: pre-dose, ½, 1, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 2-093 + Placebo
Number analyzed (Participants) | 12
hours
  tmax (BIA 2-005) | 2 [1 to 6]
  tmax (Digoxin) (Digoxin+placebo) | 1 [0.5 to 2]
  tmax (Digoxin) (Digoxin+BIA 2-093) | 1 [0.5 to 4]

3. Secondary Outcome: AUCτ - Steady-state Area Under the Plasma Concentration-time Profile Over 24 h
Description: Steady-state Area Under the Plasma Concentration-time Profile Over 24 h of BIA 2-005 (BIA 2-093 metabolite) and Digoxin
Time Frame: Day 6 and Day 7: pre-dose; Day 8: pre-dose, ½, 1, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BIA 2-093 + Placebo
Number analyzed (Participants) | 12
ng*h/mL
  AUCτ (BIA 2-005) | 370297 (79388)
  AUCτ (Digoxin) (Digoxin+Placebo) | 17607 (5599)
  AUCτ (Digoxin) (Digoxin+BIA 2-093) | 16595 (3801)

ADVERSE EVENTS:
Groups:
- BIA 2-093+Digoxin: BIA 2-093 + Digoxin
- Placebo+Digoxin: Placebo + Digoxin
Arm/Group | BIA 2-093+Digoxin | Placebo+Digoxin
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 10/13 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIA 2-093+Digoxin (N=13) | Placebo+Digoxin (N=13)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) — hypertension worsened during Period 1 (digoxin + BIA 2-093) and ameliorated during the washout;
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093+Digoxin (N=13) | Placebo+Digoxin (N=13)
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 0
Lipothymia (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 4 | 1
Somnolence (Nervous system disorders) | 3 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0
Taste bitter (Nervous system disorders) | 2 | 0
Tension headache (Nervous system disorders) | 1 | 2
Vasovagal reaction (Nervous system disorders) | 1 | 0
Axillary pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General unwell (General disorders) | 1 | 0
Retrosternal pain (General disorders) | 1 | 1
Abdominal distension & abdominal pain generalized (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Epigastric burning (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Generalized pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension worsened (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes